CLINICAL TRIAL: NCT02615470
Title: Impact of a Multicomponent Immunization Intervention on Pneumococcal and Herpes Zoster Vaccinations: A Randomized Controlled Trial of Community Pharmacies in 2 States
Brief Title: Enhancing a Sustainable Pharmacy-based Immunization Program in Two States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Keck Graduate Institute of Claremont, California (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Salisa Westrick, Professor of Health Outcomes Research and Policy, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MISP53380
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Herpes Zoster; Pneumococcal Infections
Keywords: Pneumococcal Vaccines; Shingles; Pharmacy; Vaccine; Immunization
MeSH Terms: conditions — Herpes Zoster; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced immunization delivery model (Experimental): Pharmacist-technician pairs employed by community pharmacies that are assigned to this arm will receive a) immunization update training, b) training by immunization experts to enhance immunization delivery model and foster practice change at the beginning of 6-month and c) regular feedback and clinical support for the period of 6 months.
  Interventions: Behavioral: Enhanced immunization delivery model; Other: Immunization update
- Immunization update (Active Comparator): Pharmacist-technician pairs employed by community pharmacies that are assigned to the control arm will receive an immunization update training. They will not receive a training by immunization experts nor regular feedback and clinical support.
  Interventions: Other: Immunization update

INTERVENTIONS:
Behavioral: Enhanced immunization delivery model — Webinar and online training will be delivered to intervention pharmacist-technician pairs to discuss strategies that can be used to enhance immunization delivery model and how to integrate the new model into their routine practice. This intervention also includes feedback from immunization experts for the period of 6 months.
  Arms: Enhanced immunization delivery model
Other: Immunization update — Basic immunization update online webinar will summarize changes in immunization schedules.

SUMMARY:
The study's aim is to enhance current immunization activities in community pharmacies through targeting the two most commonly available non-seasonal vaccines in community pharmacies, namely pneumococcal and herpes zoster vaccination services. The study will compare the change in the number of pneumococcal and herpes zoster vaccinations administered in pharmacy from the corresponding 6-month period prior to the intervention to the 6-month intervention period between intervention pharmacies and the control pharmacies.

DETAILED DESCRIPTION:
Community pharmacies are in a unique position and have potential to help increase immunization rates, especially among those who do not visit their primary care provider regularly. This study seeks to increase the level of pharmacy-based immunization delivery.

The study intervention is designed to increase the current level of pharmacy-based immunization delivery and foster practice change to sustain the intervention effect. Our intervention combines evidence-based strategies for improving immunization coverage and strategies to overcome system barriers to increase sustainability of the intervention over time. The study will focus on pneumococcal and herpes zoster vaccination services.

Specific aims include:

1. To compare the change in the number of pneumococcal and herpes zoster vaccinations administered in pharmacy from the corresponding 6-month period prior to the intervention to the 6-month intervention period between intervention pharmacies and the control pharmacies. The pre-intervention period will correspond to the intervention period.
2. To compare the extent of immunization activity implementation during the intervention period between intervention pharmacies and control pharmacies.
3. To compare the level of sustainability of immunization services over the period of 6 months after the intervention period ends between the intervention group and the control group.
4. To explore facilitators and barriers to implementing immunization services.
5. To explore factors affecting patient acceptance of pharmacist's vaccine recommendations within the intervention pharmacies.

ELIGIBILITY:
Inclusion Criteria:

* Alabama and California community pharmacies
* Must provide in-store prescription-dispensing service
* Must provide pneumococcal vaccine and/or herpes zoster

Exclusion Criteria:

* Must have no plan to close or change the ownership in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salisa C Westrick, PhD, Principal Investigator — Auburn University
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - Keck Graduate Institute School of Pharmacy, Claremont, California

REFERENCES:
- [Derived] Hastings TJ, Hohmann LA, Huston SA, Ha D, Westrick SC, Garza KB. Enhancing pharmacy personnel immunization-related confidence, perceived barriers, and perceived influence: The We Immunize program. J Am Pharm Assoc (2003). 2020 Mar-Apr;60(2):344-351.e2. doi: 10.1016/j.japh.2019.10.005. Epub 2019 Nov 14. PMID 31735650
- [Derived] Hohmann LA, Hastings TJ, Ha DR, Garza KB, Huston SA, Chen L, Westrick SC. Impact of a multi-component immunization intervention on pneumococcal and herpes zoster vaccinations: A randomized controlled trial of community pharmacies in 2 states. Res Social Adm Pharm. 2019 Dec;15(12):1453-1463. doi: 10.1016/j.sapharm.2019.01.006. Epub 2019 Feb 7. PMID 30777645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community pharmacies in Montgomery, Jefferson, Mobile, Tuscaloosa, Lee (AL) and San Bernadino, Riverside, Los Angeles, San Diego in CA were identified using Hayes Directory. Pharmacies were recruited via telephone with a maximum of 5 contact attempts. Eligible pharmacies must offer at least pneumococcal or herpes zoster vaccination service.
Pre-assignment Details: A randomized block design was used. Eligible community pharmacies within each block (AL and CA) were randomly assigned to each treatment group. Pharmacies with the same ownership were assigned to the same treatment group to prevent potential contamination.
Units Other Than Participants: Pharmacy
Period: Overall Study
Arm/Group | Enhanced Immunization Delivery Model | Immunization Update
Started | 58; 30 Pharmacy | 62; 32 Pharmacy
Completed the Baseline Surveys | 46; 27 Pharmacy | 47; 25 Pharmacy
Completed (Completed the 6-month survey) | 37; 22 Pharmacy | 30; 15 Pharmacy
Not Completed | 21; 8 Pharmacy | 32; 17 Pharmacy
Not completed — Lost to Follow-up | 21 | 32

BASELINE CHARACTERISTICS:
Units Other Than Participants: Pharmacy
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Immunization Delivery Model | Immunization Update | Total
Number analyzed (Participants) | 58 | 62 | 120
Number analyzed (Pharmacy) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants] — Age information was not collected per protocol specifications
  Participants
    <=18 years | NA — Age information was not collected per protocol specifications | NA — Age information was not collected per protocol specifications | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | NA — Age information was not collected per protocol specifications | NA — Age information was not collected per protocol specifications | NA — Total not calculated because data are not available (NA) in one or more arms.
    >=65 years | NA — Age information was not collected per protocol specifications | NA — Age information was not collected per protocol specifications | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data points
  Participants
    number analyzed (Participants) | 46 | 47 | 93
    Female | 34 | 29 | 63
    Male | 12 | 18 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Missing data points
  Participants
    number analyzed (Participants) | 46 | 47 | 93
    Hispanic or Latino | 4 | 5 | 9
    Not Hispanic or Latino | 38 | 40 | 78
    Unknown or Not Reported | 4 | 2 | 6
State [Count of Units; unit: Pharmacy] — State in which the pharmacies were located.
  Pharmacy
    Alabama | 17 | 18 | 35
    California | 13 | 14 | 27
Daily prescription volume [Mean (Standard Deviation); unit: prescriptions per day] — Population: The unit of analysis is pharmacy
  prescriptions per day
    number analyzed (Participants) | 46 | 47 | 93
    number analyzed (Pharmacy) | 27 | 25 | 52
    (all) | 155 (100) | 229 (124) | 192 (118)
Number of pharmacists trained in vaccine administration [Mean (Standard Deviation); unit: pharmacists] — Population: The unit of analysis is pharmacy
  pharmacists
    number analyzed (Participants) | 46 | 47 | 93
    number analyzed (Pharmacy) | 27 | 25 | 52
    (all) | 2.1 (1.5) | 2.3 (0.7) | 2.3 (1.1)
Annual pneumococcal polysaccharide (PPSV23) [Mean (Standard Deviation); unit: doses] — Self-reported vaccine dose for pneumococcal polysaccharide (PPSV23) in 2015 Population: Some pharmacies didn't provide vaccine doses
  doses
    number analyzed (Participants) | 46 | 47 | 93
    number analyzed (Pharmacy) | 27 | 25 | 52
    (all) | 7.60 (12.61) | 3.42 (5.58) | 5.56 (9.93)
Annual pneumococcal 13-valent conjugate (PCV13) [Mean (Standard Deviation); unit: doses] — Self-reported vaccine doses for pneumococcal 13-valent conjugate (PCV13) in 2015 Population: Some pharmacies didn't provide vaccine doses
  doses
    number analyzed (Participants) | 46 | 47 | 93
    number analyzed (Pharmacy) | 27 | 25 | 52
    (all) | 18.45 (26.82) | 27.16 (54.90) | 22.69 (42.51)
Annual herpes zoster [Mean (Standard Deviation); unit: doses] — Self-reported vaccine doses for herpes zoster vaccine in 2015 Population: Some pharmacies didn't provide vaccine doses
  doses
    number analyzed (Participants) | 46 | 47 | 93
    number analyzed (Pharmacy) | 27 | 25 | 52
    (all) | 14.90 (16.71) | 24.11 (28.41) | 19.38 (23.32)

OUTCOME MEASURES:

1. Primary Outcome: Number of Herpes Zoster and Pneumococcal Vaccinations Administered
Description: The change in the number of pneumococcal and herpes zoster vaccinations administered in pharmacy during the 6-month intervention period from the 6-month baseline.
Time Frame: 6 months
Population: The data was reported by the pharmacy unit; participants are part of the pharmacy unit.
Measure: Median (Inter-Quartile Range); unit: vaccine doses
Units Other Than Participants: Pharmacy
Arm/Group | Enhanced Immunization Delivery Model | Immunization Update
Number analyzed (Participants) | 37 | 30
Number analyzed (Pharmacy) | 22 | 15
vaccine doses
  Change in the total number of vaccine doses | 4.50 [-1 to 15.25] | 1 [-18 to 16]
  Change in the number of herpes zoster | 1.50 [-5 to 7] | 2 [0 to 4]
  Change in the number of pneumococcal vaccine doses | 3.5 [-.25 to 9.5] | 0 [-6 to 14]
Statistical Analysis 1: Comparison: Enhanced Immunization Delivery Model vs Immunization Update; Test type: Superiority; p = 0.202, Wilcoxon (Mann-Whitney) — A priori alpha = 0.05

2. Secondary Outcome: Number of Strategies Implemented to Promote Immunization Activities
Description: During the study, pharmacist-technician pairs engaged in on-going strategies used to advertise, market and assess non-seasonal immunization service processes. Of the total of 10 strategies possible, each pair selected strategies that they implemented. Results were reported by a representative from each pharmacy unit.
Time Frame: 6 months
Population: The unit of analysis was the pharmacy, a representative of each pharmacy unit reported the outcome. Two of the enhanced pharmacy did not provide responses regarding strategies to promote immunization activities.
Measure: Median (Inter-Quartile Range); unit: Process activities engaged
Units Other Than Participants: Pharmacy
Arm/Group | Enhanced Immunization Delivery Model | Immunization Update
Number analyzed (Participants) | 25 | 25
Number analyzed (Pharmacy) | 25 | 25
Process activities engaged | 8 [7 to 9.5] | 7 [5 to 9]
Statistical Analysis 1: Comparison: Enhanced Immunization Delivery Model vs Immunization Update; Test type: Superiority; p = 0.048, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: The Level of Sustainability of Immunization Services
Description: Change in the number of pneumococcal and herpes zoster vaccinations administered in pharmacy from 12 Months Pre- to 12 Months Post-Intervention. A representative of each pharmacy unit reported vaccine doses.
Time Frame: 24 months
Population: The unit of analysis was the pharmacy. A representative from each pharmacy unit reported the results. Results presented were collected 12 months after the intervention ended. Not all pharmacies that completed the 6 months survey completed the 12 months survey.
Measure: Median (Inter-Quartile Range); unit: vaccine doses
Units Other Than Participants: Pharmacy
Arm/Group | Enhanced Immunization Delivery Model | Immunization Update
Number analyzed (Participants) | 17 | 9
Number analyzed (Pharmacy) | 17 | 9
vaccine doses
  Change in the number of total vaccine doses | 12 [3 to 32.5] | 8 [-6 to 23.5]
  Change in the number of herpes zoster vaccine dose | 4 [-5 to 12] | 5 [-4 to 12]
  Change in the number of pneumococcal vaccine doses | 6 [1.5 to 19] | 3 [-1.5 to 19.5]
Statistical Analysis 1: Comparison: Enhanced Immunization Delivery Model vs Immunization Update; Test type: Superiority; p = 0.322, Wilcoxon (Mann-Whitney) — a priori alpha = 0.05

ADVERSE EVENTS:
Time Frame: No adverse events were monitored during the study period
Description: All cause mortality, serious adverse events and others were not monitored/assessed
Arm/Group | Enhanced Immunization Delivery Model | Immunization Update
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT02615470/Prot_SAP_000.pdf
  • Informed Consent Form (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT02615470/ICF_001.pdf